CLINICAL TRIAL: NCT00067821
Title: A Comparative Study of Pediatric CNS Tumor Activity as Assessed by 18F-FDG PET Imaging and Proton Magnetic Resonance Spectroscopic Imaging (1H-MRSI)
Brief Title: Comparison of PET and Proton MRS Imaging to Evaluate Pediatric Brain Tumor Activity
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030278; 03-C-0278; NCT00070512 (obsolete NCT alias)
Record Dates: First submitted 2003-08-28; First posted 2003-08-28 (Estimated); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Brain Tumors
Keywords: Brain Tumor; Children; Metabolic; Spectroscopy; PET; Natural History
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Patients: Must have a brain tumor, or residual abnormality that is measurable or evaluable on standard MRI or CT
  Interventions: Drug: 2-Flourodeoxyglucose

INTERVENTIONS:
Drug: 2-Flourodeoxyglucose

SUMMARY:
This study in children and young adults will compare two types of imaging, positron emission tomography ([(18)F]-DG PET) and proton magnetic resonance spectroscopy ((1)H-MRSI), to determine activity of a brain tumor or abnormal tissue in the brain following treatment for a brain tumor. Children with brain tumors are generally followed with magnetic resonance imaging (MRI) scans to evaluate response to treatment. However, because MRI only provides information on the structure of the brain, it may difficult to tell if an abnormal finding is due to tumor, swelling, scar tissue, or dead tissue. (1)H-MRSI and [(18)F]-DG PET, on the other hand, provide information on the metabolic activity of brain lesions. These two methods will be compared and evaluated for their ability to provide important additional information on childhood brain tumors.

Patients between 1 and 21 years of age with a brain tumor or brain tissue abnormality following treatment for a brain tumor may be eligible for this study. Candidates will be screened with a medical history and physical examination, pregnancy test in women who are able to become pregnant, and a blood test for glucose.

Participants will undergo the following procedures:

(1)H-MRSI - This test is similar to MRI and is done in the same scanning machine. In MRI, scans of the brain are obtained by applying a strong magnetic field and then collecting the signals released from water after the magnetic field is changed. Pictures of the brain are then obtained by computer analysis of these signals. In (1)H-MRSI, the computer blocks the signal from water to get information on brain chemicals that can indicate whether an abnormality is tumor or dead tissue. Both MRI and MRI and (1)H-MRSI are done in this study.

For these tests, the child lies on a stretcher that moves into the scanner - a narrow metal cylinder with a strong magnetic field. The child's head is placed in a headrest to prevent movement during the scan. He or she will hear loud thumping noises caused by the electrical switching of the magnetic field. A contrast agent is given through an intravenous (IV) catheter (plastic tube placed in an arm vein) or through a central line if one is in place. The contrast material brightens the images to provide a clearer picture of abnormalities. Children who have difficulty holding still or being in a scanning machine are given medications by an anesthesiologist to make them sleep through the procedure. Children who are awake during the procedure can communicate with the MRI technician at all times and ask to be removed from the scanner at any time. The MRI and (1)H-MRSI take 1-1/2 to 2 hours to complete.

[(18)F]-DG PET - For this test, [(18)F]-DG (a radioactive form of glucose) is injected into the patient's arm vein through a catheter, followed by the PET scan, similar to a very open MRI scan without the noise. The PET scan tells how active the patient's tumor is by tracking the radioactive glucose. All cells use glucose, but cells with increased metabolism, such as cancer cells, use more glucose than normal cells. After the glucose injection, the patient lies quietly in a darkened room for 30 minutes, after which he or she is asked to urinate to help reduce the dose of radiation to the bladder. Then, the scan begins. When the scan is finished (after about 1 hour), the child is asked to urinate again and then every 3 to 4 hours for the rest of the day.

Patients remain in the study for 2 years unless they withdraw, become pregnant, or require sedation but can no longer use an anesthetic. MRI and 1H-MRSI scans may be repeated every few months during the study period, if necessary. Only one PET scan is done each year.

DETAILED DESCRIPTION:
Background:

* Children with brain tumors are generally followed for response or progression by imaging studies, such as CT or MRI.
* While these imaging studies help delineate the anatomical location and extent of a tumor within the CNS, they give no information regarding the biologic or metabolic activity of the lesion.
* Proton Nuclear Magnetic Resonance Spectroscopic Imaging ((1)H-MRSI) is a non-invasive method of detecting and measuring cellular metabolites in vivo, providing biochemical information in conjunction with the spatial information obtained by MRI.
* Positron Emission Tomography (PET) is a technique that also provides data on metabolic activity of brain lesions.
* A comparison of these two methods in determining a lesion s metabolic activity has not been reported in children with brain tumors.

Objective:

-To compare (1)H-MRSI and [(18)F-]-FDG PET scanning percentage (%) of agreement between supratentorial and infratentorial tumors, and between brainstem and cerebellum intratentorial tumors.

Eligibility:

* Age: greater than or equal to 1 year and less than to 21 years
* Patients must have a brain tumor that is measurable or evaluable on standard MRI or CT.

Design:

* Patients referred for this study will have both (1)H-MRSI and (18)F-FDG PET imaging performed within 2 weeks of each other at the NCI
* Patients will remain on study for 5 years or until one of the off-study criteria have been met (whichever occurs first)

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age: greater than or equal to 1 years and less than or equal to 21 years.
  2. Radiographic diagnosis: Patients must have a brain tumor (including, but not limited to high grade gliomas, low-grade gliomas, primitive neuroectodermal tumors, ependymomas) or residual abnormality (e.g. post-operatively or post-radiation) that is measurable or evaluable on standard MRI or CT.
  3. All patients or their legal guardians (if the patient is less than 18 years of age) must sign a document of informed consent indicating their awareness of the investigational nature and the risks of this study.
  4. Prior treatment: Patients will be eligible regardless of prior treatment. Therefore, patients who are newly diagnosed, post-operative, post-radiation or post-chemotherapy are eligible.

EXCLUSION CRITERIA:

1. Patients under age 18 years who weigh greater than 70 kg are excluded because they would exceed the standard allowable dosimetry for pediatric patients (i.e. Effective Dose greater than 0.5 REM/year). In addition, patients who weigh greater than 136 kg are excluded, as this is the maximum weight allowable on PET scanner tables.
2. Pregnant or breastfeeding women
3. Any patient who is unable (either because of physical or psychological factors) to undergo imaging studies without sedation but is not considered an anesthesia candidate.
4. Any patient with a metallic MRI incompatible implant, including cardiac pacemakers, neural pacemakers, aneurysmal clips, shrapnel, cochlear implants or ferrous surgical clips.
5. Any patient with a history of a severe reaction (CTC v.4 Grade greater than or equal to 2) to Gadolinium or other contrast agents.
6. Any patient with Diabetes mellitus or steroid-induced hyperglycemia (fasting glucose greater than 150) because this may interfere with the interpretation of the [(18)F]-FDG PET scan.
7. Any patient with permanent braces, permanent retainers or nonferrous implant that, in the judgment of the Principal Investigator, would interfere with obtaining spectroscopy in the area of the tumor.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients must have a brain tumor (including, but not limited to high grade gliomas, low-grade gliomas, primitive neuroectodermal tumors, ependymomas) or residual abnormality (e.g. post-operatively or post-radiation) that is measurable or evaluable on standard MRI or CT
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Comparison | one scan each/year X 5 years
  compare results from Proton Magnetic Resonance Spectroscopic Imaging (1H-MRSI) and [18F]-FDG Positron Emission Tomography (PET) in brain tumors

SECONDARY OUTCOMES:
Evaluate change | 5 years
  To evaluate changes over time in brain tumors
Comparison | one scan each/year X 5 years
  correlate results of compare results from Proton Magnetic Resonance Spectroscopic Imaging (1H-MRSI) and [18F]-FDG Positron Emission Tomography (PET) with MRI

CONTACTS AND LOCATIONS:
Overall Officials: John W Glod, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-C-0278.html